CLINICAL TRIAL: NCT03314727
Title: Effects of Salt and The Amount of Water Consumption Simultaneously On Serum Osmolarity and Their Effects on Hemodynamic Parameters and Inflammation
Brief Title: Effects of Salt on Serum Osmolarity and Hemodynamics Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015.097.IRB2.037
Record Dates: First submitted 2017-09-28; First posted 2017-10-19 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-09

CONDITIONS: Hypertension; Sodium Excess; Oxidative Stress; Inflammation
Keywords: Osmolar Concentration; Oxidative Stress; Salt; Inflammation; Endothelial Function; Hypertension
MeSH Terms: conditions — Hypertension; Hypernatremia; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Drink 200 ml soup with no added salt
- High salt (NaCl) intake (Experimental): Group 2: Drink 200 ml soup with 3 g added salt Group 3: Drink 200 ml soup with 3 g added salt plus 500 ml water Group 4: Drink 200 ml soup with 3 g added salt plus 750 ml water
  Interventions: Other: High salt (NaCl) intake

INTERVENTIONS:
Other: High salt (NaCl) intake — Participants are asked to consume two high sodium-containing soups while monitoring their serum osmolarity levels
  Arms: High salt (NaCl) intake

SUMMARY:
Diets containing excessive salt (>12 g/day) have negative effects on kidney and cardiovascular system. Considering this known fact, the investigators aimed to study if the amount of the water taken with excessive salt had any part on these negative effects by testing the blood pressure, serum osmolality, endothelial functions, cardiac function, inflammatory parameters and sympathetic nervous system.

Excessive dietary salt raises the serum osmolality, which triggers the protection mechanisms of the body. The first mechanism is the secretion of vasopressin from posterior pituitary and the second one is the polyol mediated aldose reductase enzyme activation in renal tubules. In the beginning, water and a little amount of salt is reabsorbed from the kidneys for keeping the serum osmolality in normal ranges by the elevation of vasopressin. Besides the high levels of vasopressin for long durations may have a role in both developments of hypertension and the progression/development of chronic kidney disease. Polyol mediated aldose reductase enzyme turns glucose into sorbitol, which is turned to fructose by sorbitol dehydrogenase activity. Fructose is degraded by fructokinase activity into toxic substances. With this pathway, the acute energy need is satisfied, yet uric acid, local oxidative stress, and inflammatory mediators rise while nitric oxide levels decreasing. These facts are independent risk factors for both kidney disease progression and hypertension. In addition, excessive salt intake may elevate the transforming growth factor beta-1 (TGF-B1) levels, which activates the sympathetic system, inflammation, and endothelial dysfunction.

According to these data, the investigators speculate that if they increase the amount of water intake while eating the high salt diet they may decrease the toxic effect of salt with less increase in serum osmolarity. To test this hypothesis, by regulating the salt and water amount in healthy people's diets, the investigators aimed to evaluate the following these parameters; biochemical parameters that could affect the blood and urine osmolality, blood pressure, vascular endothelial functions with the non-invasive flow-mediated dilatation technique and arterial stiffness, systolic and diastolic functions of the heart by transthoracic echocardiography. In addition, it was planned to evaluate the hormonal effects of arginine vasopressin, a long peptide with 39 amino acids, which is longer and easier to measure than vasopressin levels in serum by measuring the pituitary hormone-derived copeptin.

Although, decreasing the salt intake is the first step of the treatment in hypertension, and kidney diseases, the compliance rate to less sodium intake is very low (<20%). The investigators aim is to evaluate the effects of water, which is taken acutely with the excessive salt intake on cardiovascular system and kidney. The findings of the study will important for public health. If the investigators prove their hypothesis, they may recommend increasing high water intake before feeling thirst of which may contribute to decreasing the prevalence of hypertension and kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, no smoker, no obese >30 BMI, no drug use in the previous month

Exclusion Criteria:

* Any systemic disease, no past history of any cardiovascular disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline systolic and diastolic blood pressure | Baseline time 0, Hour 1, Hour 2, Hour 3, Hour 4
  Systolic and diastolic blood pressures are measured with an aneroid sphygmomanometer. Unit of measurement is mmHg.

SECONDARY OUTCOMES:
Serum osmolarity increase | Baseline time 0, Hour 1, Hour 2, Hour 3, Hour 4
  2x[Na]+[Glucose]/18+[Blood Urea Nitrogen]/2.8
Change from baseline blood copeptin levels | Baseline time 0, Hour 1, Hour 2, Hour 3, Hour 4
  Blood concentration in pg/ml
Change from baseline augmentation index | Baseline time 0, Hour 4
  Augmentation index (AIx@75) is the difference between the second and the first peaks of the central aortic waveform expressed as the percentage (%) of the aortic pulse pressure. It is measured non invasively using Mobil Pulse Wave Analysis device from brachial artery. This outcome measure will be used for the assessment of arterial stiffness.
Change from baseline pulse wave velocity | Baseline time 0, Hour 4
  Pulse wave velocity (PWV) is the travel time (m/s) of a pressure wave from common carotid to the brachial artery, as a measure of aortic compliance. It is measured non invasively using Mobil Pulse Wave Analysis device from brachial artery. This outcome measure will be used for the assessment of arterial stiffness.
Change from baseline flow mediated dilation | Baseline time 0, Hour 4
  Endothelial function was measured via noninvasive ultrasound imaging. Participants were asked to lie supine for a 10-minute resting period where a three-lead ECG was placed for monitoring of heart rate and rhythm throughout the procedures. Standard ultrasonography equipment (Epiq 7, Philips Medical, and Bothell, WA) with a 12-megahertz linear array probe was used to obtain B-mode images of the left brachial artery approximately 2-10 cm proximal to the elbow. Following measurement of resting artery diameter, a blood pressure cuff was placed distally to the brachial artery (antecubital space) and inflated to a suprasystolic level (200 mm/Hg) for 5 minutes to induce ischemia. After the abrupt release of the cuff pressure, changes in blood flow and vessel diameter (FMD) over a 5-minute period were imaged.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kanbay, MD, Principal Investigator — Koc University Sch. Med. Dept. Internal Med. Nephrology
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)